CLINICAL TRIAL: NCT01511497
Title: A Randomized, Placebo Controlled, Double-Blind, Third Party Open, Ascending Dose Study To Evaluate The Safety, Tolerability, Pharmacokinetics And Pharmacodynamics Of PF-04427429 Administered Intravenously To Healthy Female Adult Volunteers
Brief Title: Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics Study Of PF-04427429 In Healthy Women Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B0141008
Record Dates: First submitted 2011-10-18; First posted 2012-01-18 (Estimated); Last update posted 2013-02-21 (Estimated); Status verified 2013-02

CONDITIONS: Pain; Migraine Disorders
Keywords: Phase 1; PF-04427429
MeSH Terms: conditions — Pain; Migraine Disorders | interventions — Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- PF-04427429 (Experimental)
  Interventions: Biological: PF-04427429
- Placebo (Placebo Comparator): Normal saline
  Interventions: Other: Normal saline

INTERVENTIONS:
Biological: PF-04427429 — Intravenous, single dose given over 1 hour with experimental dose. Subjects can receive one of four potential doses - 300, 1000, 1500 or 2000 mg.
  Arms: PF-04427429
Other: Normal saline — Intravenous, normal saline
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the safety, tolerability, pharmacokinetics, and pharmacodynamics of PF-04427429 in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Generally healthy women, of non-child bearing potential, between the ages of 18 and 65 years, inclusive. Healthy is defined as no clinically relevant abnormalities identified by a detailed medical history, full physical examination, including blood pressure and pulse rate measurement, 12-lead ECG or clinical laboratory tests.
* Body Mass Index (BMI) of 17.5 to 35.0 kg/m2; and a total body weight between 50 kg (110 lbs) and 120 kg (265 lbs) inclusive.

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, hepatic, psychiatric, or neurologic, disease. Subjects with asymptomatic, seasonal allergies at the time of dosing will not be excluded.
* Women of childbearing potential.
* History or diagnosis of ocular disease or conditions that would confound the assessment of ocular safety, such as diabetic retinopathy, uveitis, severe wet or dry AMD.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2011-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Screening up to Day 168
Incidence and severity of clinical laboratory abnormalities. | Screening up to Day 168
Mean change from baseline and placebo in blood pressure (BP). | Screening up to Day 168
Mean change from baseline in 12-lead electrocardiogram (ECG) parameters compared to baseline and placebo. | Screening up to Day 168
Categorical summary of QTcF compared to baseline between dose groups and placebo. | Screening up to Day 168
Anti-Drug Antibodies (ADA) responses. | From Day 0 up to Day 168 and until levels return to baseline.
Intravenous (IV) injection site reactions. | Day 1 post dose
Mean change from baseline and placebo in pulse rate (PR). | Screening up to Day 168
Mean change from baseline and placebo in body temperature. | Screening up to Day 168

SECONDARY OUTCOMES:
Area under the concentration-time curve from zero to infinite time postdose (AUCinf). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Time to maximum concentration (Tmax). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Maximum concentration (Cmax). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Area under the concentration-time curve from zero to the last quantifiable concentration (AUClast). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Terminal elimination half-life (t½). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Clearance (CL). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168
Volume of distribution (Vz). | Days 1, 2, 3, 4, 7, 14, 28, 42, 56, 70, 84 & 168

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Dallas, Texas

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=B0141008&StudyName=Safety%2C%20Tolerability%2C%20Pharmacokinetics%2C%20and%20Pharmacodynamics%20Study%20Of%20PF-04427429%20In%20Healthy%20Women%20Volunteers